CLINICAL TRIAL: NCT05168800
Title: CONFIDENT: A Randomized Trial to Increase COVID-19 Vaccine Confidence in Long-term Care Workers
Brief Title: CONFIDENT: Supporting Long-term Care Workers During COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Association of Health Care Assistants (Unknown); Institute for Healthcare Improvement (Other); East Carolina University (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Glyn Jones-Elwyn, Professor, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00032340
Record Dates: First submitted 2021-12-21; First posted 2021-12-23 (Actual); Results first posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dialogue-Based Webinar (Experimental)
  Interventions: Behavioral: Dialogue-Based Webinar
- Social Media Website (Experimental)
  Interventions: Behavioral: Social Media Website
- Enhanced Usual Practice (Active Comparator)
  Interventions: Other: Enhanced Usual Practice

INTERVENTIONS:
Behavioral: Dialogue-Based Webinar — One-time virtual webinars facilitated by a long-term care worker and a physician expert. The webinars will include provision of the existing COVID-19 vaccine Option Grid(TM) conversation aid. The majority of time will be focused on answering participants' questions about COVID-19 and the COVID-19 vaccines. An additional refresher intervention will be delivered several weeks later that will comprise of an email with links to a pre-recorded, shorter webinar available in video and audio-only formats.
  Other Names: Discussion Session
  Arms: Dialogue-Based Webinar
Behavioral: Social Media Website — A curated COVID-19 social media website. The website will feature content from different social media platforms. The posts will include information about COVID-19 and the COVID-19 vaccines. Participants will have the ability to like and comment on website content and can re-visit the website as many times as they like. An additional refresher intervention will be delivered several weeks later that will comprise of an email featuring previews and links to a selection of website content.
  Other Names: Social Site
  Arms: Social Media Website
Other: Enhanced Usual Practice — COVID-19 vaccine information on the Centers for Disease Control and Prevention (CDC) website. An additional refresher will be delivered several weeks later that will comprise of an email with a link to the COVID-19 vaccine information on the CDC website.
  Other Names: Online Information
  Arms: Enhanced Usual Practice

SUMMARY:
The CONFIDENT Study is an online three-arm randomized trial that aims to help long-term care workers in the United States feel more confident about the Coronavirus Disease 2019 (COVID-19) vaccines. The study will compare two different interventions to usual online information (website of the Centers for Disease Control and Prevention). The first intervention is a Dialogue-Based Webinar where people can interact and ask questions about the vaccines. The second intervention is a Social Media Website that will feature curated content about the vaccines from popular social media platforms.

Participants will be asked to completed four online surveys. The first survey will be completed pre-intervention and immediately upon study enrollment (Time 0). Participants will be randomized to a trial arm at the end of the Time 0 survey. Intervention follow-up surveys will be completed 3 weeks post-randomization (Time 1), three months post-randomization (Time 2), and 6 months post-randomization (Time 3).

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* can read, write, and understand English
* lives in the United States
* has worked in a long-term care setting in the past two years
* can provide information to confirm they have worked in a long-term care setting
* is not pregnant or breastfeeding
* at least somewhat worried about the COVID-19 vaccines and/or has not received a COVID-19 vaccine booster shot

Exclusion Criteria:

* under 18 years of age
* cannot read, write, and understand English
* does not live in the United States
* has not worked in a long-term care setting in the past two years
* cannot provide information to confirm they have worked in a long-term care setting
* is pregnant or breastfeeding
* less than somewhat worried about the COVID-19 vaccines and has received at least one COVID-19 vaccine booster shot

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2634 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glyn Elwyn, Principal Investigator — Dartmouth College
Locations (1):
- Dartmouth College, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified copy of participant-level data and essential analytic code will be made available to others for research purposes, via data sharing.
Supporting Information: Study Protocol, SAP, Analytic Code

REFERENCES:
- [Background] Larson HJ, de Figueiredo A, Xiahong Z, Schulz WS, Verger P, Johnston IG, Cook AR, Jones NS. The State of Vaccine Confidence 2016: Global Insights Through a 67-Country Survey. EBioMedicine. 2016 Oct;12:295-301. doi: 10.1016/j.ebiom.2016.08.042. Epub 2016 Sep 13. PMID 27658738
- [Background] Hamel L, Lopes L, Kirzinger A, Sparks G, Stokes M, Brodie M. KFF COVID-19 Vaccine Monitor: Media and Misinformation. 2021 Nov. Available at: https://www.kff.org/coronavirus-covid-19/poll-finding/kff-covid-19-vaccine-monitor-media-and-misinformation/
- [Derived] Stevens G, Johnson LC, Saunders CH, Schmidt P, Sierpe A, Thomeer RP, Little NR, Cantrell M, Yen RW, Pogue JA, Holahan T, Schubbe DC, Forcino RC, Fillbrook B, Sheppard R, Wooten C, Goldmann D, O'Malley AJ, Dube E, Durand MA, Elwyn G. The CONFIDENT study protocol: a randomized controlled trial comparing two methods to increase long-term care worker confidence in the COVID-19 vaccines. BMC Public Health. 2023 Feb 23;23(1):384. doi: 10.1186/s12889-023-15266-x. PMID 36823559

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was initially launched on February 21, 2022. After nearly three weeks of recruitment, we experienced a large amount of fraudulent study enrollment and had to pause recruitment for a period of time. We relaunched the study on May 5, 2022. No data from the initial launch was used in data analyses given differences in study eligibility, participant verification processes, and time that had elapsed between the two groups. For more details, see: https://pubmed.ncbi.nlm.nih.gov/38588798/
Pre-assignment Details: A total of 14,984 people were screened for eligibility. Randomization occurred automatically at the end of the study baseline survey (Time 0). Pre-randomization exclusions were as follows: did not meet inclusion criteria (n=9,285); did not consent (n=1,354); dropped out of survey before randomization (n=1,711). Post-randomization exclusions are detailed in the Participant Flow.
Period: Time 1 Survey
Arm/Group | Dialogue-Based Webinar | Social Media Website | Enhanced Usual Practice
Started (Completed baseline survey (Time 0) and randomized to a trial arm) | 877 | 878 | 879
Completed (In final Time 1 sample) | 426 | 474 | 487
Not Completed | 451 | 404 | 392
Not completed — Did not start T1 survey | 182 | 150 | 140
Not completed — Completed T1 survey outside window | 18 | 21 | 13
Not completed — Missing primary outcome data at Time 0 or Time 1 | 1 | 6 | 1
Not completed — Failed verification, did not start Time 1 survey | 221 | 200 | 220
Not completed — Failed verification, did complete time 1 survey | 23 | 24 | 16
Not completed — Withdrawal by Subject | 6 | 3 | 2
Period: Time 2 Survey
Arm/Group | Dialogue-Based Webinar | Social Media Website | Enhanced Usual Practice
Started (Invited to Time 2 survey) | 654 | 676 | 660
Completed (In final Time 2 sample) | 384 | 432 | 431
Not Completed | 270 | 244 | 229
Not completed — Already excluded at Time 1 | 228 | 202 | 173
Not completed — Did not start Time 2 survey | 31 | 26 | 45
Not completed — Completed Time 2 survey outside window | 10 | 15 | 9
Not completed — Missing primary outcome data at Time 2 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1
Period: Time 3 Survey
Arm/Group | Dialogue-Based Webinar | Social Media Website | Enhanced Usual Practice
Started (Invited to Time 3 survey) | 653 | 674 | 659
Completed (In final Time 3 sample) | 376 | 419 | 427
Not Completed | 277 | 255 | 232
Not completed — Already excluded at Time 1 | 228 | 200 | 173
Not completed — Did not start Time 3 survey | 48 | 48 | 51
Not completed — Completed Time 3 survey outside window | 1 | 6 | 8
Not completed — Missing primary outcome data at Time 3 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Overall number of baseline participants is calculated based on the final sample used for primary outcome analyses at Time 1.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dialogue-Based Webinar | Social Media Website | Enhanced Usual Practice | Total
Number analyzed (Participants) | 426 | 474 | 487 | 1387
Age, Customized [Count of Participants; unit: Participants]
  Under age 50 | 364 | 401 | 400 | 1165
  Age 50-64 | 56 | 71 | 80 | 207
  Age 65 and older | 6 | 2 | 7 | 15
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 399 | 451 | 464 | 1314
  Male | 24 | 22 | 21 | 67
  Nonbinary or preferred to self-describe | 3 | 1 | 2 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White non-hispanic | 260 | 300 | 292 | 852
  Black non-hispanic | 124 | 120 | 131 | 375
  Hispanic | 19 | 23 | 27 | 69
  Other race or more than one race | 22 | 30 | 35 | 87
  Missing | 1 | 1 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: COVID-19 Vaccine Confidence
Description: Confidence in the COVID-19 vaccines, assessed using the 3-item Vaccine Confidence Index (Larson et al., 2016) adapted for COVID-19. Each item is rated on a 5-point scale ranging from 1 ('Strongly disagree') to 5 ('Strongly agree'). Respondents are considered 'confident' (score of '1') if they respond 'Agree' or 'Strongly agree' on all three items and 'not confident' (score of '0') if one or more item responses is not 'Agree' or 'Strongly agree'.
Time Frame: 3 weeks post-randomization (Time 1)
Measure: Count of Participants; unit: Participants
Arm/Group | Dialogue-Based Webinar | Social Media Website | Enhanced Usual Practice
Number analyzed (Participants) | 426 | 474 | 487
Participants | 93 | 106 | 138
Statistical Analysis 1: Comparison: Dialogue-Based Webinar vs Enhanced Usual Practice; Test type: Superiority; p = 0.99, Groupwise binomial comparison — To achieve a group-wise 95% confidence for the primary outcome, each of the three tests were evaluated with acceptance based on a 98.4% confidence interval, or greater than 2.15 standard deviations of the mean for the superiority analyses
Statistical Analysis 2: Comparison: Social Media Website vs Enhanced Usual Practice; Test type: Superiority; p = 0.98, Groupwise binomial comparison — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Dialogue-Based Webinar vs Social Media Website; Test type: Equivalence — A sample size of 1800 LTCWs (600 per arm) was identified to provide 80% power to detect an 8% difference in the rate of individuals reporting vaccine confidence between arms with 95% confidence. This sample size was sufficient to retain 80% power to detect a 10% difference after 40% attrition. Per study design, the equivalence margin is +/- 10% with anticipated attrition using the binomial confidence interval; p = 0.85, Groupwise binomial comparison — To achieve a group-wise 95% confidence for the primary outcome, each of the three tests were evaluated with acceptance based on a 98.4% confidence interval, or +/- 2.45 standard deviations of the mean for the equivalency test

2. Secondary Outcome: Change From Baseline to 3 Weeks Post-randomization in COVID-19 Vaccine Confidence
Description: Change in confidence in the COVID-19 vaccines from baseline to 3 weeks post-randomization, assessed using the 3-item Vaccine Confidence Index (Larson et al., 2016) adapted for COVID-19. Each item is rated on a 5-point scale ranging from 1 ('Strongly disagree') to 5 ('Strongly agree'). Respondents are considered 'confident' (score of '1') if they respond 'Agree' or 'Strongly agree' on all three items and 'not confident' (score of '0') if one or more item responses is not 'Agree' or 'Strongly agree'. For the change from baseline to Time 1 outcome, a score of 1 represents an increase in vaccine confidence (Vaccine Confidence Index score change from 0 to 1) and a score of 0 represents no change or a decrease in confidence.
Time Frame: Baseline (Time 0); 3 weeks post-randomization (Time 1)
Measure: Count of Participants; unit: Participants
Arm/Group | Dialogue-Based Webinar | Social Media Website | Enhanced Usual Practice
Number analyzed (Participants) | 426 | 474 | 487
Participants | 42 | 49 | 62
Statistical Analysis 1: Comparison: Dialogue-Based Webinar vs Enhanced Usual Practice; Test type: Superiority; p = 0.93, Fisher Exact
Statistical Analysis 2: Comparison: Social Media Website vs Enhanced Usual Practice; Test type: Superiority; p = 0.90, Fisher Exact
Statistical Analysis 3: Comparison: Dialogue-Based Webinar vs Social Media Website; Test type: Equivalence — The study was not powered for secondary outcome analyses; p = 0.83, Fisher Exact

3. Secondary Outcome: Change From Baseline to 3 Months Post-randomization in COVID-19 Vaccine Confidence
Description: Change in confidence in the COVID-19 vaccines from baseline to 3 months post-randomization, assessed using the 3-item Vaccine Confidence Index (Larson et al., 2016) adapted for COVID-19. Each item is rated on a 5-point scale ranging from 1 ('Strongly disagree') to 5 ('Strongly agree'). Respondents are considered 'confident' (score of '1') if they respond 'Agree' or 'Strongly agree' on all three items and 'not confident' (score of '0') if one or more item responses is not 'Agree' or 'Strongly agree'. For the change from baseline to Time 2 outcome, a score of 1 represents an increase in vaccine confidence (Vaccine Confidence Index score change from 0 to 1) and a score of 0 represents no change or a decrease in confidence.
Time Frame: Baseline (Time 0); 3 months post-randomization (Time 2)
Population: Number of participants analyzed is less than the Time 1 analyzed sample due to participants either not completing the Time 2 survey and/or the vaccine confidence survey questions.
Measure: Count of Participants; unit: Participants
Arm/Group | Dialogue-Based Webinar | Social Media Website | Enhanced Usual Practice
Number analyzed (Participants) | 384 | 432 | 431
Participants | 57 | 58 | 55
Statistical Analysis 1: Comparison: Dialogue-Based Webinar vs Enhanced Usual Practice; Test type: Superiority; p = 0.22, Fisher Exact
Statistical Analysis 2: Comparison: Social Media Website vs Enhanced Usual Practice; Test type: Superiority; p = 0.43, Fisher Exact
Statistical Analysis 3: Comparison: Dialogue-Based Webinar vs Social Media Website; Test type: Equivalence — The study was not powered for secondary outcome analyses; p = 0.61, Fisher Exact

4. Secondary Outcome: Change From Baseline to 6 Months Post-randomization in COVID-19 Vaccine Confidence
Description: Change in confidence in the COVID-19 vaccines from baseline to 6 months post-randomization, assessed using the 3-item Vaccine Confidence Index (Larson et al., 2016) adapted for COVID-19. Each item is rated on a 5-point scale ranging from 1 ('Strongly disagree') to 5 ('Strongly agree'). Respondents are considered 'confident' (score of '1') if they respond 'Agree' or 'Strongly agree' on all three items and 'not confident' (score of '0') if one or more item responses is not 'Agree' or 'Strongly agree'. For the change from baseline to Time 3 outcome, a score of 1 represents an increase in vaccine confidence (Vaccine Confidence Index score change from 0 to 1) and a score of 0 represents no change or a decrease in confidence.
Time Frame: Baseline (Time 0); 6 months post-randomization (Time 3)
Population: Number of participants analyzed is less than the Time 1 analyzed sample due to participants either not completing the Time 3 survey and/or the vaccine confidence survey questions.
Measure: Count of Participants; unit: Participants
Arm/Group | Dialogue-Based Webinar | Social Media Website | Enhanced Usual Practice
Number analyzed (Participants) | 376 | 419 | 427
Participants | 52 | 66 | 62
Statistical Analysis 1: Comparison: Dialogue-Based Webinar vs Enhanced Usual Practice; Test type: Superiority; p = 0.65, Fisher Exact
Statistical Analysis 2: Comparison: Social Media Website vs Enhanced Usual Practice; Test type: Superiority; p = 0.34, Fisher Exact
Statistical Analysis 3: Comparison: Dialogue-Based Webinar vs Social Media Website; Test type: Equivalence — The study was not powered for secondary outcome analyses; p = 0.48, Fisher Exact

5. Secondary Outcome: Net Promoter Score (COVID-19 Vaccination)
Description: Likelihood of recommending COVID-19 vaccination to someone who is not vaccinated, assessed using a single-item adapted Net Promoter Score item. The item is assessed on an 11-point scale ranging from 0 ('No at all likely') to 10 ('Extremely likely'). Responses are categorized into three groups: Promoters (scale score of 9 or 10) receive a score of '1', passives (scale score of 7 or 8) receive a score of '0', and detractors (scale score of 0-6) receive a score of '-1'.
Time Frame: 3 weeks post-randomization (Time 1)
Population: Arm totals do not equal overall baseline analysis population due to missing data (i.e., unanswered survey questions).
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Dialogue-Based Webinar | Social Media Website | Enhanced Usual Practice
Number analyzed (Participants) | 421 | 462 | 477
score on a scale | -0.48 (0.04) | -0.52 (0.03) | -0.42 (0.04)
Statistical Analysis 1: Comparison: Dialogue-Based Webinar vs Enhanced Usual Practice; Test type: Superiority; p = 0.88, Adjusted Wald test
Statistical Analysis 2: Comparison: Social Media Website vs Enhanced Usual Practice; Test type: Superiority; p = 0.97, Adjusted Wald test
Statistical Analysis 3: Comparison: Dialogue-Based Webinar vs Social Media Website; Test type: Equivalence — The study was not powered for secondary outcome analyses; p = 0.48, Adjusted Wald test

6. Secondary Outcome: Net Promoter Score (COVID-19 Booster Vaccination to Coworker)
Description: Likelihood of recommending COVID-19 booster vaccination to a coworker, assessed using a single-item adapted Net Promoter Score item. The item is assessed on an 11-point scale ranging from 0 ('No at all likely') to 10 ('Extremely likely'). Responses are categorized into three groups: Promoters (scale score of 9 or 10) receive a score of '1', passives (scale score of 7 or 8) receive a score of '0', and detractors (scale score of 0-6) receive a score of '-1'.
Time Frame: 3 weeks post-randomization (Time 1)
Population: Arm totals do not equal overall baseline analysis population due to missing data (i.e., unanswered survey questions).
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Dialogue-Based Webinar | Social Media Website | Enhanced Usual Practice
Number analyzed (Participants) | 421 | 467 | 481
score on a scale | -0.59 (0.09) | -0.62 (0.04) | -0.51 (0.04)
Statistical Analysis 1: Comparison: Dialogue-Based Webinar vs Enhanced Usual Practice; Test type: Superiority; p = 0.95, Adjusted Wald test
Statistical Analysis 2: Comparison: Social Media Website vs Enhanced Usual Practice; Test type: Superiority; p = 0.98, Adjusted Wald test
Statistical Analysis 3: Comparison: Dialogue-Based Webinar vs Social Media Website; Test type: Equivalence — The study was not powered for secondary outcome analyses; p = 0.66, Adjusted Wald test

7. Secondary Outcome: COVID-19 Vaccine Uptake (Any Dose)
Description: Receipt of any does of a COVID-19 vaccine, assessed using a single item with multiple choice (single answer) format.
Time Frame: 3 weeks post-randomization (Time 1)
Measure: Count of Participants; unit: Participants
Arm/Group | Dialogue-Based Webinar | Social Media Website | Enhanced Usual Practice
Number analyzed (Participants) | 426 | 474 | 487
Participants | 363 | 383 | 397
Statistical Analysis 1: Comparison: Dialogue-Based Webinar vs Enhanced Usual Practice; Test type: Superiority; p = 0.08, Fisher Exact
Statistical Analysis 2: Comparison: Social Media Website vs Enhanced Usual Practice; Test type: Superiority; p = 0.64, Fisher Exact
Statistical Analysis 3: Comparison: Dialogue-Based Webinar vs Social Media Website; Test type: Equivalence — The study was not powered for secondary outcome analyses; p = 0.09, Fisher Exact

8. Secondary Outcome: COVID-19 Vaccine Uptake (Initial Series Completion)
Description: Completion of initial COVID-19 vaccine series, assessed using two items with multiple choice (single answer) formats.
Time Frame: 3 weeks post-randomization (Time 1)
Measure: Count of Participants; unit: Participants
Arm/Group | Dialogue-Based Webinar | Social Media Website | Enhanced Usual Practice
Number analyzed (Participants) | 426 | 474 | 487
Participants | 354 | 374 | 391
Statistical Analysis 1: Comparison: Dialogue-Based Webinar vs Enhanced Usual Practice; Test type: Superiority; p = 0.13, Fisher Exact
Statistical Analysis 2: Comparison: Social Media Website vs Enhanced Usual Practice; Test type: Superiority; p = 0.73, Fisher Exact
Statistical Analysis 3: Comparison: Dialogue-Based Webinar vs Social Media Website; Test type: Equivalence — The study was not powered for secondary outcome analyses; p = 0.10, Fisher Exact

9. Secondary Outcome: COVID-19 Vaccine Uptake (Booster Completion)
Description: Receipt of a COVID-19 booster vaccine if initial series completed, assessed using a single item with multiple choice (single answer) format.
Time Frame: 3 weeks post-randomization (Time 1)
Measure: Count of Participants; unit: Participants
Arm/Group | Dialogue-Based Webinar | Social Media Website | Enhanced Usual Practice
Number analyzed (Participants) | 426 | 474 | 487
Participants | 132 | 144 | 145
Statistical Analysis 1: Comparison: Dialogue-Based Webinar vs Enhanced Usual Practice; Test type: Superiority; p = 0.37, Fisher Exact
Statistical Analysis 2: Comparison: Social Media Website vs Enhanced Usual Practice; Test type: Superiority; p = 0.45, Fisher Exact
Statistical Analysis 3: Comparison: Dialogue-Based Webinar vs Social Media Website; Test type: Equivalence — The study was not powered for secondary outcome analyses; p = 0.88, Fisher Exact

10. Secondary Outcome: COVID-19 Vaccine Intent (Initial Series)
Description: Intent to get a COVID-19 vaccine if unvaccinated, assessed using a single item with multiple choice (single answer) format. Response options are Yes (score of '1'), Not Sure (score of '0'), and No (score of '-1').
Time Frame: 3 weeks post-randomization (Time 1)
Population: Only participants who reported not having received any dose of a COVID-19 vaccine at Time 1 received this question, therefore, arm totals do not equal overall baseline analysis population.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Dialogue-Based Webinar | Social Media Website | Enhanced Usual Practice
Number analyzed (Participants) | 63 | 91 | 89
score on a scale | -0.76 (0.07) | -0.77 (0.05) | -0.62 (0.06)
Statistical Analysis 1: Comparison: Dialogue-Based Webinar vs Enhanced Usual Practice; Test type: Superiority; p = 0.92, Adjusted Wald test
Statistical Analysis 2: Comparison: Social Media Website vs Enhanced Usual Practice; Test type: Superiority; p = 0.97, Adjusted Wald test
Statistical Analysis 3: Comparison: Dialogue-Based Webinar vs Social Media Website; Test type: Equivalence — The study was not powered for secondary outcome analyses; p = 0.83, Adjusted Wald test

11. Secondary Outcome: COVID-19 Vaccine Intent (Booster)
Description: Intent to get a COVID-19 booster vaccine if not yet received, assessed using a single item with multiple choice (single answer) format. Response options are Yes (score of '1'), Not Sure (score of '0'), and No (score of '-1').
Time Frame: 3 weeks post-randomization (Time 1)
Population: Only participants who reported completing their initial vaccine series but not having received a COVID-19 booster vaccine at Time 1 received this question, therefore, arm totals do not equal overall baseline analysis population.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Dialogue-Based Webinar | Social Media Website | Enhanced Usual Practice
Number analyzed (Participants) | 212 | 219 | 240
score on a scale | -0.26 (0.05) | -0.16 (0.05) | -0.17 (0.05)
Statistical Analysis 1: Comparison: Dialogue-Based Webinar vs Enhanced Usual Practice; Test type: Superiority; p = 0.88, Adjusted Wald test
Statistical Analysis 2: Comparison: Social Media Website vs Enhanced Usual Practice; Test type: Superiority; p = 0.49, Adjusted Wald test
Statistical Analysis 3: Comparison: Dialogue-Based Webinar vs Social Media Website; Test type: Equivalence — The study was not powered for secondary outcome analyses; p = 0.23, Adjusted Wald test

12. Secondary Outcome: COVID-19 Vaccine Intent (Future Vaccine Recommendations)
Description: Intent to get COVID-19 vaccines regularly in the future if they are recommended, assessed using a single item with multiple choice (single answer) format. Response options are Yes (score of '1'), Not Sure (score of '0'), and No (score of '-1').
Time Frame: 3 weeks post-randomization (Time 1)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Dialogue-Based Webinar | Social Media Website | Enhanced Usual Practice
Number analyzed (Participants) | 426 | 474 | 487
score on a scale | -0.16 (0.04) | -0.17 (0.04) | -0.09 (0.04)
Statistical Analysis 1: Comparison: Dialogue-Based Webinar vs Enhanced Usual Practice; Test type: Superiority; p = 0.90, Adjusted Wald test
Statistical Analysis 2: Comparison: Social Media Website vs Enhanced Usual Practice; Test type: Superiority; p = 0.94, Adjusted Wald test
Statistical Analysis 3: Comparison: Dialogue-Based Webinar vs Social Media Website; Test type: Equivalence — The study was not powered for secondary outcome analyses; p = 0.86, Adjusted Wald test

13. Secondary Outcome: Feeling Informed About the COVID-19 Vaccines
Description: Extent of feeling informed (having enough information and understanding that information) about the COVID-19 vaccines, using two self-developed items. Each item is assessed on a 5-point scale ranging from 0 ('No at all confident') to 4 ('Very confident'). A single overall score is calculated as the mean of the two items (possible range 0-4).
Time Frame: 3 weeks post-randomization (Time 1)
Population: Arm totals do not equal overall baseline analysis population due to missing data (i.e., unanswered survey questions).
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Dialogue-Based Webinar | Social Media Website | Enhanced Usual Practice
Number analyzed (Participants) | 414 | 466 | 481
score on a scale | 2.68 (0.05) | 2.68 (0.05) | 2.89 (0.05)
Statistical Analysis 1: Comparison: Dialogue-Based Webinar vs Enhanced Usual Practice; Test type: Superiority; p = 1.00, Two-sample z test
Statistical Analysis 2: Comparison: Social Media Website vs Enhanced Usual Practice; Test type: Superiority; p = 1.0, Two-sample z test
Statistical Analysis 3: Comparison: Dialogue-Based Webinar vs Social Media Website; Test type: Equivalence — The study was not powered for secondary outcome analyses; p = 0.49, Two-sample z test

14. Secondary Outcome: Identification of COVID-19 Vaccine Information and Misinformation
Description: Identification of COVID-19 vaccine information and misinformation, assessed using four items. Some items self-developed and some adapted from Hamel et al., 2021. Each item is assessed using a multiple choice (single answer) format. Each item response is scored as correct (value of '1') or incorrect (value of '0'). A single overall score is calculated as the sum of all four items (possible range 0-4).
Time Frame: 3 weeks post-randomization (Time 1)
Population: Social media website arm total does not equal overall baseline analysis population due to one case of missing data (i.e., unanswered survey question/s).
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Dialogue-Based Webinar | Social Media Website | Enhanced Usual Practice
Number analyzed (Participants) | 426 | 473 | 487
score on a scale | 2.19 (0.07) | 2.00 (0.06) | 2.30 (0.06)
Statistical Analysis 1: Comparison: Dialogue-Based Webinar vs Enhanced Usual Practice; Test type: Superiority; p = 0.88, Two-sample z test
Statistical Analysis 2: Comparison: Social Media Website vs Enhanced Usual Practice; Test type: Superiority; p = 1.00, Two-sample z test
Statistical Analysis 3: Comparison: Dialogue-Based Webinar vs Social Media Website; Test type: Equivalence — The study was not powered for secondary outcome analyses; p = 0.02, Two-sample z test

15. Secondary Outcome: Trust in COVID-19 Vaccine Information From Different Sources
Description: Trust in COVID-19 vaccine information given by different people and organizations, assessed using a list of three different sources. Each source is assessed using a 4-point scale ranging from 0 ('Not at all') to 3 ('A lot'). A single overall score is calculated as the mean of the three items (possible range 0-3).
Time Frame: 3 weeks post-randomization (Time 1)
Population: Arm totals do not equal overall baseline analysis population due to missing data (i.e., unanswered survey questions).
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Dialogue-Based Webinar | Social Media Website | Enhanced Usual Practice
Number analyzed (Participants) | 424 | 471 | 485
score on a scale | 1.71 (0.05) | 1.65 (0.04) | 1.76 (0.04)
Statistical Analysis 1: Comparison: Dialogue-Based Webinar vs Enhanced Usual Practice; Test type: Superiority; p = 0.82, Two-sample z test
Statistical Analysis 2: Comparison: Social Media Website vs Enhanced Usual Practice; Test type: Superiority; p = 0.97, Two-sample z test
Statistical Analysis 3: Comparison: Dialogue-Based Webinar vs Social Media Website; Test type: Equivalence — The study was not powered for secondary outcome analyses; p = 0.18, Two-sample z test

16. Secondary Outcome: Change From Baseline in Secondary Outcomes
Description: Change in secondary outcomes from baseline, assessed using the same measures identified in Outcomes 3-13.
Time Frame: Baseline (Time 0); 3 weeks post-randomization (Time 1); 3 months post-randomization (Time 2); 6 months post-randomization (Time 3)
Reporting Status: Not Posted

17. Secondary Outcome: As-treated Analyses of Primary and Secondary Outcomes
Description: All primary and secondary outcomes assessed only for those who were exposed to their relevant study intervention and/or refresher intervention.
Time Frame: as for outcome 16
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Dialogue-Based Webinar Exposure
Description: Participants' exposure to the Dialogue-Based Webinar intervention assessed via webinar attendance data.
Time Frame: Time of individual participants' exposure to intervention
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Social Media Website Exposure
Description: Participants' exposure to the Social Media Website intervention assessed via website visit data.
Time Frame: Time of individual participants' exposure to intervention
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Dialogue-Based Webinar Acceptability
Description: Likelihood of recommending the Dialogue-Based Webinar intervention to a coworker, assessed using a single-item adapted Net Promoter Score item.
Time Frame: 3 weeks post-randomization (Time 1); 3 months post-randomization (Time 2)
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Social Media Website Acceptability
Description: Likelihood of recommending the Social Media Website intervention to a coworker, assessed using a single-item adapted Net Promoter Score item.
Time Frame: 3 weeks post-randomization (Time 1); 3 months post-randomization (Time 2)
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Enhanced Usual Practice Acceptability
Description: Likelihood of recommending the Centers for Disease Control and Prevention (CDC) website to a coworker, assessed using a single-item adapted Net Promoter Score item.
Time Frame: 3 weeks post-randomization (Time 1); 3 months post-randomization (Time 2)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Each participant was monitored for adverse events per their trial arm. Webinar and Usual Practice arms: participants were monitored from Time 0 survey completion to completion of their last survey (maximum of approx. 6 months duration for each participant). Website arm: participants were monitored from Time 0 survey completion to when the Website was closed on September 20, 2023. Monitoring in this arm for each participant ranged from approx. 8-19 months depending on when they joined the study.
Arm/Group | Dialogue-Based Webinar | Social Media Website | Enhanced Usual Practice
All-Cause Mortality (participants affected / at risk) | 0/426 | 0/474 | 0/487
Serious Adverse Events (participants affected / at risk) | 0/426 | 0/474 | 0/487
Other Adverse Events (participants affected / at risk) | 0/426 | 0/474 | 0/487

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-08): https://cdn.clinicaltrials.gov/large-docs/00/NCT05168800/Prot_SAP_000.pdf